CLINICAL TRIAL: NCT04627363
Title: HAIC Synchronously Combined With Bevacizumab and Toripalimab First-line for Advanced Hepatocellular Carcinama
Brief Title: HAIC Combined With Bevacizumab and Toripalimab for Advanced Hepatocellular Carcinama
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYEYJR-3
Record Dates: First submitted 2020-11-12; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Hepatocellular Carcinoma; Bevacizumab; Liver Neoplasms; Toripalimab; Oxaliplatin
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Bevacizumab; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC plus Bevacizumab and Toripalimab (Experimental): Hepatic arterial infusion of oxaliplatin , fluorouracil, and leucovorin every 6 weeks. Lenvatinib 12 mg (or 8 mg) once daily (QD) oral dosing. Toripalimab, 240 mg intravenously every 3 weeks. Bevacizumab 15 mg/kg intravenously every 3 weeks.
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Bevacizumab; Drug: Toripalimab

INTERVENTIONS:
Procedure: Hepatic arterial infusion chemotherapy — administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries every 6 weeks
Drug: Bevacizumab — 15mg/kg intravenously every 3 weeks
Drug: Toripalimab — 240mg intravenously every 3 weeks

SUMMARY:
This is an open-label, single-arm clinical study to preliminarily observe and evaluate the efficacy and safety of hepatic arterial infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin synchronous combined with Bevacizumab and Toripalimab as the first-line therapy for advanced HCC.

DETAILED DESCRIPTION:
Hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin, 5-fluorouracil and leucovorin was effective and safe for hepatocellular carcinoma. Bevacizumab, an angiogenesis Inhibitors was effectively used for hepatocelluar carcinama (HCC) therapy. Toripalimab, an programmed cell death protein-1 (PD-1) antibody, was effective and tolerable in patients with hepatocellular carcinoma and portal vein tumor thrombus. No study has evaluated HAIC plus Bevacizumab and Toripalimab. Thus, the investigators carried out this prospective, single-arm study to find out it.

ELIGIBILITY:
Inclusion Criteria:

1. HCC diagnosed by histopathological examination or Guidelines for Diagnosis and Treatment of Primary Liver Cancer or the recurrent HCC after surgery;
2. age between 18 and 75 years;
3. Stage B (middle stage) or C (late stage) HCC determined in accordance with Barcelona Clinic Liver Cancer staging system (BCLC stage). In case of stage B.
4. No previous use of any systemic therapy or recurrent HCC.
5. Child-Pugh class A or B;
6. Eastern Cooperative Group performance status (ECOG) score of 0-2;
7. Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3
8. Prothrombin time ≤18s or international normalized ratio < 1.7.
9. Ability to understand the protocol and to agree to and sign a written informed consent document.

Exclusion Criteria:

1. Cholangiocellular carcinoma (ICC);
2. Patients with cancer thrombus in the main trunk of portal vein (Vp4), or cancer thrombus in inferior vena cava should be excluded;
3. Accepting ablation or surgery or other system therapy as firt line therapy after diagnose for primary HCC, ablation or system therapy as first line therapy for recurrent HCC.
4. Serious medical comorbidities.
5. Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
6. Known history of HIV
7. History of organ allograft
8. Known or suspected allergy to the investigational agents or any agent given in association with this trial.
9. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
10. Evidence of bleeding diathesis.
11. Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rate at 6 months | 6 months]
  Progression was defined as progressive disease by independent radiologic review according to mRECIST or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 6 months
  OS is the length of time from the date of randomization until death from any cause.
Progression free survival (PFS) | 6 months
  PFS is defined as the time from the date of randomization to the date of the first objectively documented tumor progression or death due to any cause.
Objective response rate (ORR) | 6 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all randomized subjects whose best overall response (BOR) is either a CR or PR.
Adverse events | 6 months
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Gao, Study Director — Sun Yat-sen University; Kangshun Zhu, Professor, Study Director — Second Affiliated Hospital of Guangzhou Medical University

IPD SHARING:
Plan to Share IPD: No